CLINICAL TRIAL: NCT05174000
Title: An Open-label, Single-dose, Randomized, 4-period, 2-sequence, Fully Replicated Crossover, Single-center Phase I Study to Assess Bioequivalence in Healthy Participants Between Euthyrox® Tablets Manufactured at Merck Nantong Versus Euthyrox® Tablets Manufactured at Merck Darmstadt Administered Orally as 12 Tablets of 50 μg
Brief Title: BE of Euthyrox® Tablets (Merck Nantong Versus Merck Darmstadt Sites)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200125_0006
Record Dates: First submitted 2021-12-20; First posted 2021-12-30 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Euthyrox®; Bioequivalence; Thyroid-Stimulating Hormone; Thyroxine
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1:Test Euthyrox®, then Reference Euthyrox®, then Test Euthyrox®, then Reference Euthyrox® (Experimental): Participants will receive single oral dose of Test Euthyrox® on in treatment period 1, followed by single oral dose of Reference Euthyrox® in treatment period 2, followed by single oral dose of Test Euthyrox® in treatment period 3, followed by single oral dose of Reference Euthyrox in treatment period 4. Participants will remain resident until Day 4 for each treatment period and there will be a washout period of 53 days between each treatment period.
  Interventions: Drug: Test Euthyrox®; Drug: Reference Euthyrox®
- Sequence 2:Reference Euthyrox®, then Test Euthyrox®, then Reference Euthyrox®, then Test Euthyrox® (Experimental): Participants will receive single oral dose of Reference Euthyrox® in treatment period 1, followed by single oral dose of Test Euthyrox® in treatment period 2, followed by single oral dose of Reference Euthyrox® in treatment period 3, followed by single oral dose of Test Euthyrox® in treatment period 4. Participants will remain resident until Day 4 for each treatment period and there will be a washout period of 53 days between each treatment period.
  Interventions: Drug: Test Euthyrox®; Drug: Reference Euthyrox®

INTERVENTIONS:
Drug: Test Euthyrox® — Participants will receive single oral dose of Test Euthyrox® either in treatment period 1, 2, 3 or 4.
  Other Names: Levothyroxine sodium
Drug: Reference Euthyrox® — Participants will receive single oral dose of Reference Euthyrox® either in treatment period 1, 2, 3 or 4.
  Other Names: Levothyroxine sodium

SUMMARY:
The purpose of this study is to demonstrate bioequivalence (BE) between Euthyrox® tablets manufactured at Merck Nantong (Test Euthyrox) versus the tablets manufactured at Merck Darmstadt (Reference Euthyrox).

ELIGIBILITY:
Inclusion Criteria:

* Participants have a body weight within 45 to 75 kilogram (kg) for females and 55 to 85 kg for males and Body mass index (BMI) within the range 19.0 to 26.0 kilograms per meter square (kg/m^2)
* Non-smoker for at least 3 months
* Contraceptive use by males or females will be consistent with any local regulations on contraception methods for those participating in clinical studies
* Capable of giving signed informed consent
* Total and free Thyroxine (T4), total and free Triiodothyronine (T3) and Thyroid-stimulating Hormone (TSH) must be within normal ranges at Screening
* Ability to understand the purposes and risks of the study
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history or presence of tumors of the pituitary gland or hypothalamus, thyroid or adrenal gland dysfunction or cardiac disease
* Participants with a concurrent medical condition known to interfere with the absorption or metabolism of thyroid hormones
* History or presence of relevant liver diseases or hepatic dysfunction. Participants with gall bladder removal
* Participants taking medications known to affect thyroid hormone metabolism, for example, oral contraceptives, hormonal implants, parenteral hormones, anabolic steroids, androgens, etcetera
* Use of any investigational device within 60 days prior to first dose administration
* Pregnant or breastfeeding a child
* Participant has smoked within the 3 months prior to Screening
* High fiber consumption within 24 hours before dosing in each period
* Participants with positive results from serology examination for Syphilis, Hepatitis B surface antigen, Hepatitis C Virus or Human Immunodeficiency Virus
* Participants with any clinically relevant abnormality in the safety laboratory parameters
* Participants with positive test for drugs of abuse (including alcohol) at Screening and on Day -1 of each period (urine)
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration, Adjusted for Baseline (Cmax[adj]) of Total Thyroxine (T4) | Pre-dose up to 72 hours post-dose
Baseline-Corrected Area Under the Serum Concentration-Time Curve (AUC) from Time Zero to 72 hours Post-dose (AUC0-72,adj) of Total Thyroxine (T4) | Pre-dose up to 72 hours post-dose

SECONDARY OUTCOMES:
Serum Concentrations of Total Thyroxine (T4) and Triiodothyronine (T3) | Pre-dose up to 72 hours post-dose
Safety Profile as Assessed by Occurrence of Severity of Treatment-emergent Adverse Events (TEAEs), Laboratory Variables, Vital Signs and 12-Lead Electrocardiogram (ECG) Measurements | Baseline up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200125_0006
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html